CLINICAL TRIAL: NCT03126110
Title: A Phase 1/2 Study Exploring the Safety, Tolerability, and Efficacy of INCAGN01876 in Combination With Immune Therapies in Subjects With Advanced or Metastatic Malignancies
Brief Title: Phase 1/2 Study Exploring the Safety, Tolerability, and Efficacy of INCAGN01876 Combined With Immune Therapies in Advanced or Metastatic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCAGN 1876-201; 2016-004989-25 (EudraCT Number)
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Results first posted 2022-12-28 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced Malignancies; Metastatic Cancer
Keywords: cervical cancer; endometrial cancer; gastric cancer (stomach, esophageal, and gastroesophageal junction [GEJ]); hepatocellular carcinoma (HCC); melanoma; Merkel cell carcinoma; mesothelioma; microsatellite instability-high (MSI-H) colorectal cancer (CRC); non-small cell lung cancer (NSCLC); ovarian cancer; squamous cell carcinoma of the head and neck (SCCHN); small cell lung cancer (SCLC); renal cell carcinoma (RCC); triple-negative breast cancer (TNBC); urothelial carcinoma; glucocorticoid-induced tumor necrosis factor receptor (GITR)
MeSH Terms: conditions — Neoplasm Metastasis; Uterine Cervical Neoplasms; Endometrial Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Melanoma; Carcinoma, Merkel Cell; Mesothelioma; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Squamous Cell Carcinoma of Head and Neck; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + nivolumab 240 mg Q2W (Experimental): Participants received INCAGN01876 1.0 milligrams per kilogram (mg/kg) administered intravenously (IV) every 2 weeks (Q2W) in combination with nivolumab 240 mg administered IV Q2W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + nivolumab 240 mg Q2W (Experimental): Participants received INCAGN01876 3.0 mg/kg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + nivolumab 240 mg Q2W (Experimental): Participants received INCAGN01876 5.0 mg/kg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + nivolumab 240 mg Q2W (Experimental): Participants received INCAGN01876 10.0 mg/kg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, then nivolumab 240 mg Q2W (Experimental): Participants received INCAGN01876 1.0 mg/kg administered IV Q2W for a total of 2 doses as run-in, followed by INCAGN01876 1.0 mg/kg Q2W in combination with nivolumab 240 mg administered IV Q2W starting at Cycle 3.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, then nivolumab 240 mg Q2W (Experimental): Participants received INCAGN01876 1.0 mg/kg administered IV Q2W for a total of 2 doses as run-in, followed by INCAGN01876 1.0 mg/kg Q2W in combination with nivolumab 240 mg administered IV Q2W starting at Cycle 3.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, then nivolumab 240 mg Q2W (Experimental): Participants received INCAGN01876 5.0 mg/kg administered IV Q2W for a total of 2 doses as run-in, followed by INCAGN01876 5.0 mg/kg Q2W in combination with nivolumab 240 mg administered IV Q2W starting at Cycle 3.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + ipilimumab 1 mg/kg Q6W (Experimental): Participants received INCAGN01876 1.0 mg/kg administered IV Q2W in combination with ipilimumab 1 mg/kg administered IV every 6 weeks (Q6W).
  Interventions: Drug: INCAGN01876; Drug: Ipilimumab
- Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + ipilimumab 1 mg/kg Q6W (Experimental): Participants received INCAGN01876 3.0 mg/kg administered IV Q2W in combination with ipilimumab 1 mg/kg administered IV Q6W.
  Interventions: Drug: INCAGN01876; Drug: Ipilimumab
- Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + ipilimumab 1 mg/kg Q6W (Experimental): Participants received INCAGN01876 5.0 mg/kg administered IV Q2W in combination with ipilimumab 1 mg/kg administered IV Q6W.
  Interventions: Drug: INCAGN01876; Drug: Ipilimumab
- Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab (Experimental): Participants received INCAGN01876 1.0 mg/kg administered IV Q2W in combination with nivolumab 3 mg/kg administered IV Q2W and ipilimumab 1 mg/kg administered IV Q6W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab; Drug: Ipilimumab
- Phase 2 Group C2 PD-1/PD-L1: INCAGN01876 300 mg + ipilimumab 1 mg/kg (Experimental): Participants with programmed cell death protein/programmed cell death ligand 1 (PD-1/PD-L1) relapsed melanoma received INCAGN01876 300 mg administered IV Q2W in combination with ipilimumab 1 mg/kg administered IV Q6W.
  Interventions: Drug: INCAGN01876; Drug: Ipilimumab
- Phase 2 Group F GC: INCAGN01876 300 mg + nivolumab 240 mg (Experimental): Participants with gastric cancer (GC) received INCAGN01876 300 mg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 2 Group F SCCHN INCAGN01876 300 mg + nivolumab 240 mg (Experimental): Participants with squamous cell carcinoma of the head and neck (SCCHN) received INCAGN01876 300 mg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 2 Group F CC: INCAGN01876 300 mg + nivolumab 240 mg (Experimental): Participants with cervical cancer (CC) received INCAGN01876 300 mg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 2 Group F PD-1/PD-L1: INCAGN01876 300 mg + nivolumab 240 mg (Experimental): Participants with PD-1/PD-L1 relapsed melanoma received INCAGN01876 300 mg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab
- Phase 2 Group F Biopsy: INCAGN01876 300 mg + nivolumab 240 mg (Experimental): Participants with gastric cancer, squamous cell carcinoma of the head and neck, cervical cancer, or PD-1/PD-L1 relapsed melanoma who had tumor lesions that were amenable to percutaneous biopsy received INCAGN01876 300 mg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
  Interventions: Drug: INCAGN01876; Drug: Nivolumab

INTERVENTIONS:
Drug: INCAGN01876 — In Phase 1 participants will receive INCAGN01876 administered intravenously (IV) at the protocol-defined dose according to cohort enrollment. In Phase 2, participants will be administered IV study drug at the recommended dose from Phase 1 ().
Drug: Nivolumab — Nivolumab will be administered IV at the protocol-defined dose according to assigned treatment group.
  Arms: Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + nivolumab 240 mg Q2W; Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + nivolumab 240 mg Q2W; Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + nivolumab 240 mg Q2W; Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + nivolumab 240 mg Q2W; Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, then nivolumab 240 mg Q2W; Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, then nivolumab 240 mg Q2W; Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, then nivolumab 240 mg Q2W; Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab; Phase 2 Group F Biopsy: INCAGN01876 300 mg + nivolumab 240 mg; Phase 2 Group F CC: INCAGN01876 300 mg + nivolumab 240 mg; Phase 2 Group F GC: INCAGN01876 300 mg + nivolumab 240 mg; Phase 2 Group F PD-1/PD-L1: INCAGN01876 300 mg + nivolumab 240 mg; Phase 2 Group F SCCHN INCAGN01876 300 mg + nivolumab 240 mg
Drug: Ipilimumab — Ipilimumab will be administered IV at the protocol-defined dose according to assigned treatment group.
  Arms: Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + ipilimumab 1 mg/kg Q6W; Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + ipilimumab 1 mg/kg Q6W; Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + ipilimumab 1 mg/kg Q6W; Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab; Phase 2 Group C2 PD-1/PD-L1: INCAGN01876 300 mg + ipilimumab 1 mg/kg

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and efficacy of INCAGN01876 when given in combination with immune therapies in subjects with advanced or metastatic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent.
* Phase 1: Subjects with advanced or metastatic solid tumors.
* Phase 1: Subjects who have disease progression after treatment with available therapies.
* Phase 2: Subjects with advanced or metastatic cervical cancer, gastric cancer (including stomach, esophageal, and GEJ), SCCHN, PD-1 refractory SCCHN and PD-1/PD-L1 relapsed melanoma.
* Presence of measurable disease based on RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.

Exclusion Criteria:

* Laboratory and medical history parameters not within the Protocol-defined range
* Prior treatment with any tumor necrosis factor super family agonist.
* Receipt of anticancer medications or investigational drugs within protocol-defined intervals before the first administration of study drug.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy.
* Active autoimmune disease.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Evidence of active, noninfectious pneumonitis or history of interstitial lung disease.
* Evidence of hepatitis B virus or hepatitis C virus infection or risk of reactivation.
* Known history of human immunodeficiency virus (HIV; HIV 1/2 antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Janik, MD, Study Director — Incyte Corporation
Locations (38):
- United States (15):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University - Siteman Cancer Center, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Oklahoma, Sarah Cannon Research Institute, Oklahoma City, Oklahoma
  - Providance Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Sarah Cannon Research Institute, Nashville, Tennessee
  - BUMC Mary Crowley Cancer Research Centers, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (5):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Scientia Clinical Research, Randwick, New South Wales
  - Greenslopes Private Hospital, Brisbane, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Linear Clinical Research, Perth, Western Australia
- Belgium (8):
  - CHA Centre Hospitalier de l'Ardenne, Libramont, Chevigny
  - Saint Augustinus Hospital, Antwerp
  - Institut Jules Bordet, Brussels
  - CHU Brugmann, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Mi Kryviy Rih Center of Dnipropetrovsk Regional Council, Charleroi
  - Ghent University Hospital, Ghent
  - AZ Groeninge, Kortrijk
- Spain (10):
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Clinico y Provincial de Barcelona, Barcelona
  - Institut Catala D'Oncologia-Badalona, Barcelona
  - Hospital Vall de Hebron, Barcelona
  - Hospital Reina Sophia, Córdoba
  - University Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital HM Sanchinarro, Madrid
  - Clinica Universidad De Navarra (CUN), Pamplona
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 32 study centers in Australia, Belgium, Spain, and the United States.
Groups:
- Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W: Participants received INCAGN01876 1.0 mg/kg administered IV Q2W for a total of 2 doses as run-in, followed by nivolumab 240 mg administered IV Q2W starting at Cycle 3.
- Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W: Participants received INCAGN01876 3.0 mg/kg administered IV Q2W for a total of 2 doses as run-in, followed by nivolumab 240 mg administered IV Q2W starting at Cycle 3.
- Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W: Participants received INCAGN01876 5.0 mg/kg administered IV Q2W for a total of 2 doses as run-in, followed by nivolumab 240 mg administered IV Q2W starting at Cycle 3.
- Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg: Participants with programmed cell death protein/programmed cell death ligand 1 (PD-1/PD-L1) relapsed melanoma (RM) received INCAGN01876 300 mg administered IV Q2W in combination with ipilimumab 1 mg/kg administered IV Q6W.
- Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg: Participants with PD-1/PD-L1 relapsed melanoma received INCAGN01876 300 mg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
Period: Phase 1
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Started | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 5 | 4 | 5 | 4 | 3 | 4 | 8 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 4 | 3 | 4 | 4 | 3 | 4 | 5 | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Safety follow-up no longer necessary | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Survival follow-up no longer necessary | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 16 | 46 | 18 | 4 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 16 | 34 | 16 | 4 | 2
Not completed — Study terminated by the sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 12 | 25 | 11 | 3 | 2
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Started new treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants enrolled in the study who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg | Total
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6 | 8 | 16 | 46 | 18 | 4 | 2 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (7.37) | 59.8 (14.03) | 48.0 (18.23) | 62.3 (7.04) | 60.8 (12.40) | 62.5 (16.36) | 63.0 (9.90) | 61.5 (11.73) | 61.8 (7.70) | 67.7 (4.16) | 58.5 (11.24) | 69.1 (9.46) | 59.1 (10.48) | 60.5 (9.46) | 48.6 (9.43) | 54.3 (9.29) | 42.0 (16.97) | 58.56 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 3 | 3 | 3 | 3 | 3 | 5 | 1 | 2 | 3 | 5 | 8 | 18 | 1 | 1 | 68
  Male | 2 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 3 | 2 | 4 | 5 | 11 | 38 | 0 | 3 | 1 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 8
  Not Hispanic or Latino | 3 | 3 | 4 | 4 | 4 | 4 | 4 | 4 | 7 | 3 | 6 | 8 | 14 | 43 | 17 | 4 | 2 | 134
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 3
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    White/Caucasian | 2 | 3 | 4 | 3 | 2 | 3 | 4 | 3 | 6 | 3 | 6 | 8 | 14 | 45 | 16 | 4 | 2 | 128
    Black or African American | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 7
    Asian | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiin or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Other: Captured as "Other" | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    Other: Zimbabwean | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Other: Mexican | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study medication.
Time Frame: up to approximately 27.4 months
Population: Phase 1 Full Analysis Set (FAS): all participants enrolled in Phase 1 of the study who received at least 1 dose of INCAGN01876, nivolumab, or ipilimumab
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W: Participants received INCAGN01876 1.0 mg/kg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
- Phase 1 Group D: INCAGN01876 1.0 mg/kg + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg: Participants received INCAGN01876 1.0 mg/kg administered IV Q2W in combination with nivolumab 3 mg/kg administered IV Q2W and ipilimumab 1 mg/kg administered IV Q6W.
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 1.0 mg/kg + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6
Participants | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 7 | 3 | 6

2. Primary Outcome: Phase 2: Objective Response Rate (ORR) Per RECIST v1.1
Description: ORR was defined as the percentage of participants with a best overall response of confirmed complete response (CR) or partial response (PR), determined by investigator assessment of radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1). CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to approximately 44.7 months
Population: Phase 2 Response Evaluable Population: all participants enrolled in Phase 2 who received at least 1 dose of INCAGN01876, nivolumab, or ipilimumab; completed a Baseline scan; and met at least 1 of the following criteria: (a) ≥1 post-Baseline scan (b) the participant has been in the study for a minimum of 64 days of follow-up; or (c) the participant had discontinued from treatment
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 8 | 16 | 46 | 18 | 4 | 2
Percentage of Participants | 0.0 | 0.0 | 23.9 | 16.7 | 0.0 | 0.0

3. Secondary Outcome: Phase 1: ORR Per RECIST v1.1
Description: ORR was defined as the percentage of participants with a best overall response of unconfirmed CR or PR, determined by investigator assessment of radiographic disease assessments per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to approximately 44.7 months
Population: Phase 1 Response Evaluable Population: all participants enrolled in Phase 1 who received at least 1 dose of INCAGN01876, nivolumab, or ipilimumab; completed a Baseline scan; and met at least 1 of the following criteria: (a) ≥1 post-Baseline scan (b) the participant has been in the study for a minimum of 64 days of follow-up; or (c) the participant had discontinued from treatment
Measure: Number; unit: Percentage of Participants
Groups:
- Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W: Participants received INCAGN01876 1.0 milligrams per kilogram (mg/kg) administered intravenously (IV) every 2 weeks (Q2W) in combination with nivolumab 240 mg administered IV Q2W.INCAGN01876 combined with nivolumab.
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6
Percentage of Participants | 25.0 | 0.0 | 20.0 | 0.0 | 0.0 | 0.0 | 25.0 | 25.0 | 12.5 | 0.0 | 0.0

4. Secondary Outcome: Phase 1: ORR Per Modified RECIST (mRECIST) v1.1
Description: ORR was defined as the percentage of participants with a best overall response of unconfirmed CR or PR, determined by investigator assessment of radiographic disease assessments per mRECIST v1.1. The response of target lesions was evaluated from the percentage change in the sum of the diameters of the viable portions (portions enhanced during the arterial phase). CR: Disappearance of any intratumoral arterial enhancement during in target lesions, disappearance of all non-target lesions, and no appearance of any new lesions. PR: ≥30% of the sum of the diameters of viable portions (enhancement on arterial phase) of target lesions taking as reference the Baseline sum, no new lesions, and no progression of non-target lesions.
Time Frame: up to approximately 44.7 months
Population: Phase 1 Response Evaluable Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6
Percentage of Participants | 25.0 | 0.0 | 20.0 | 0.0 | 0.0 | 0.0 | 25.0 | 25.0 | 12.5 | 0.0 | 0.0

5. Secondary Outcome: Phase 2: ORR Per mRECIST v1.1
Description: ORR was defined as the percentage of participants with a best overall response of confirmed CR or PR, determined by investigator assessment of radiographic disease assessments per mRECIST v1.1. The response of target lesions was evaluated from the percentage change in the sum of the diameters of the viable portions (portions enhanced during the arterial phase). CR: Disappearance of any intratumoral arterial enhancement during in target lesions, disappearance of all non-target lesions, and no appearance of any new lesions. PR: ≥30% of the sum of the diameters of viable portions (enhancement on arterial phase) of target lesions taking as reference the Baseline sum, no new lesions, and no progression of non-target lesions.
Time Frame: up to approximately 44.7 months
Population: Phase 2 Response Evaluable Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 8 | 16 | 46 | 18 | 4 | 2
Percentage of Participants | 0.0 | 0.0 | 26.1 | 16.7 | 0.0 | 0.0

6. Secondary Outcome: Phase 1: Duration of Response (DOR) Per RECIST v1.1
Description: DOR was defined as the time from the first overall response contributing to an unconfirmed objective response (CR or PR) to the earlier of the participant's death from any cause or the first assessment of PD, determined by investigator assessment of radiographic disease assessment per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to approximately 44.7 months
Population: Phase 1 Response Evaluable Population. Only those participants with a response of CR or PR were analyzed. The confidence interval for median survival time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |  | 573.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |  |  |  | 876.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 281.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |  |

7. Secondary Outcome: Phase 2: DOR Per RECIST v1.1
Description: DOR was defined as the time from the first overall response contributing to a confirmed objective response (CR or PR) to the earlier of the participant's death from any cause or the first assessment of PD, determined by investigator assessment of radiographic disease assessment per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to approximately 44.7 months
Population: Phase 2 Response Evaluable Population. Only those participants with a response of CR or PR were analyzed. The confidence interval for median survival time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Phase 2 Group C2: PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg: Participants with programmed cell death protein/programmed cell death ligand 1 (PD-1/PD-L1) relapsed melanoma (RM) received INCAGN01876 300 mg administered IV Q2W in combination with ipilimumab 1 mg/kg administered IV Q6W.
- Phase 2 Group F: Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg: Participants with gastric cancer, squamous cell carcinoma of the head and neck, cervical cancer, or PD-1/PD-L1 relapsed melanoma who had tumor lesions that were amenable to percutaneous biopsy received INCAGN01876 300 mg administered IV Q2W in combination with nivolumab 240 mg administered IV Q2W.
Arm/Group | Phase 2 Group C2: PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F: Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 0 | 0 | 11 | 3 | 0 | 0
Days |  |  | NA [118.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 120.0 [113.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. |  |

8. Secondary Outcome: Phase 1: DOR Per mRECIST v1.1
Description: DOR was defined as the time from the first unconfirmed overall response contributing to an unconfirmed objective response (CR or PR) to the earlier of the participant's death from any cause or the first confirmed assessment of PD, determined by investigator assessment of radiographic disease assessment per mRECIST v1.1. The response of target lesions was evaluated from the percentage change in the sum of the diameters of the viable portions (portions enhanced during the arterial phase). CR: Disappearance of any intratumoral arterial enhancement during in target lesions, disappearance of all non-target lesions, and no appearance of any new lesions. PR: ≥30% of the sum of the diameters of viable portions (enhancement on arterial phase) of target lesions taking as reference the Baseline sum, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to approximately 44.7 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 1.0 mg/kg + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |  | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |  |  |  | 876.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |  |

9. Secondary Outcome: Phase 2: DOR Per mRECIST v1.1
Description: DOR was defined as the time from the first overall response contributing to a confirmed objective response (CR or PR) to the earlier of the participant's death from any cause or the first assessment of PD, determined by investigator assessment of radiographic disease assessment per mRECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to approximately 44.7 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2 Group C2: PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F: Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 0 | 0 | 12 | 3 | 0 | 0
Days |  |  | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [113.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. |  |

10. Secondary Outcome: Phase 1: Disease Control Rate (DCR) Per RECIST v1.1
Description: DCR was defined as the percentage of participants with a best overall response of unconfirmed CR, unconfirmed PR, or stable disease (SD; ≥49 days), determined by investigator assessment of radiographic disease assessments per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to approximately 44.7 months
Population: Phase 1 Response Evaluable Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 1.0 mg/kg + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6
Percentage of Participants | 25.0 | 50.0 | 20.0 | 50.0 | 0.0 | 25.0 | 50.0 | 25.0 | 50.0 | 0.0 | 0.0

11. Secondary Outcome: Phase 2: DCR Per RECIST v1.1
Description: DCR was defined as the percentage of participants with a best overall response of confirmed CR, confirmed PR, or SD (≥49 days), determined by investigator assessment of radiographic disease assessments per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to approximately 44.7 months
Population: Phase 2 Response Evaluable Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2 Group C2: PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F: Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 8 | 16 | 46 | 18 | 4 | 2
Percentage of Participants | 37.5 | 56.3 | 54.3 | 55.6 | 50.0 | 50.0

12. Secondary Outcome: Phase 1: DCR Per mRECIST v1.1
Description: as for outcome 10
Time Frame: up to approximately 44.7 months
Population: Phase 1 Response Evaluable Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 1.0 mg/kg + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6
Percentage of Participants | 25.0 | 50.0 | 20.0 | 50.0 | 0.0 | 25.0 | 50.0 | 25.0 | 50.0 | 0.0 | 0.0

13. Secondary Outcome: Phase 2: DCR Per mRECIST v1.1
Description: DCR was defined as the percentage of participants with a best overall response of confirmed CR, confirmed PR, or SD (≥49 days), determined by investigator assessment of radiographic disease assessments per mRECIST v1.1. The response of target lesions was evaluated from the percentage change in the sum of the diameters of the viable portions (portions enhanced during the arterial phase). CR: Disappearance of any intratumoral arterial enhancement during in target lesions, disappearance of all non-target lesions, and no appearance of any new lesions. PR: ≥30% of the sum of the diameters of viable portions (enhancement on arterial phase) of target lesions taking as reference the Baseline sum, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to approximately 44.7 months
Population: Phase 2 Response Evaluable Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2 Group C2: PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F: Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 8 | 16 | 46 | 18 | 4 | 2
Percentage of Participants | 37.5 | 56.3 | 56.5 | 55.6 | 50.0 | 50.0

14. Secondary Outcome: Phase 1: Duration of Disease Control Per RECIST v1.1
Description: Duration of disease control (CR, PR, and SD [≥49 days]) was measured from the start of treatment until PD or death from any cause, if occurring sooner than progression, determined by investigator assessment of radiographic disease per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to approximately 44.7 months
Population: Phase 1 Response Evaluable Population. The confidence intervals was calculated based on the exact method for binomial distributions. Only those participants with a response of SD, CR, or PR were analyzed.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 1.0 mg/kg + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 2 | 1 | 2 | 0 | 1 | 2 | 1 | 4 | 0 | 0
Days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [89.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 624.0 [NA to NA] — The median was not estimable because too few participants had disease progression or died. | 76.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |  | 167.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 668.5 [125.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 250.5 [110.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. |  |

15. Secondary Outcome: Phase 2: Duration of Disease Control Per RECIST v1.1
Description: as for outcome 14
Time Frame: up to approximately 44.7 months
Population: Phase 2 Response Evaluable Population. The confidence intervals was calculated based on the exact method for binomial distributions. Only those participants with a response of SD, CR, or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2 Group C2: PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F: Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 3 | 9 | 25 | 10 | 2 | 1
Days | 218.0 [106.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 109.0 [63.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 253.0 [156.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 168.0 [71.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 206.5 [118.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 109.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died.

16. Secondary Outcome: Phase 1: Duration of Disease Control Per mRECIST v1.1
Description: Duration of disease control (CR, PR, and SD [≥49 days]) was measured from the start of treatment until PD or death from any cause, if occurring sooner than progression, determined by investigator assessment of radiographic disease per RECIST v1.1. The response of target lesions was evaluated from the percentage change in the sum of the diameters of the viable portions (portions enhanced during the arterial phase). CR: Disappearance of any intratumoral arterial enhancement during in target lesions, disappearance of all non-target lesions, and no appearance of any new lesions. PR: ≥30% of the sum of the diameters of viable portions (enhancement on arterial phase) of target lesions taking as reference the Baseline sum, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to approximately 44.7 months
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 1.0 mg/kg + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 2 | 1 | 2 | 0 | 1 | 2 | 1 | 4 | 0 | 0
Days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 76.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |  | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 668.5 [125.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [134.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. |  |

17. Secondary Outcome: Phase 2: Duration of Disease Control Per mRECIST v1.1
Description: Duration of disease control (CR, PR, and SD [≥49 days]) was measured from the start of treatment until PD or death from any cause, if occurring sooner than progression, determined by investigator assessment of radiographic disease per RECIST v1.1. The response of target lesions was evaluated from the percentage change in the sum of the diameters of the viable portions (portions enhanced during the arterial phase). CR: Disappearance of any intratumoral arterial enhancement during in target lesions, disappearance of all non-target lesions, and no appearance of any new lesions. PR: ≥30% of the sum of the diameters of viable portions (enhancement on arterial phase) of target lesions taking as reference the Baseline sum, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD. [
Time Frame: up to approximately 44.7 months
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2 Group C2: PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F: Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 3 | 9 | 26 | 10 | 2 | 1
Days | 218.0 [133.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 168.0 [63.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | NA [202.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | NA [137.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | NA [118.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died.

18. Secondary Outcome: Phase 1: Progression-free Survival (PFS) Per RECIST v1.1
Description: According to RECIST 1.1, PFS was defined as the length of time between the Baseline visit (Day 1) and the earlier of death or the first assessment of PD, as determined by investigator assessment of objective radiographic disease assessments.
Time Frame: up to approximately 44.7 months
Population: Phase 1 FAS. Median survival time was estimated using the Kaplan-Meier method. The confidence interval for median survival time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6
Days | 52.5 [48.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 72.0 [53.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 53.0 [9.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 64.0 [48.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 47.5 [29.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 60.0 [50.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 88.5 [44.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 41.0 [15.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 110.0 [53.0 to 276.0] | 56.0 [53.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 54.5 [21.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

19. Secondary Outcome: Phase 2: PFS Per RECIST v1.1
Description: as for outcome 18
Time Frame: up to approximately 44.7 months
Population: Phase 2 FAS. Median survival time was estimated using the Kaplan-Meier method. The confidence interval for median survival time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 8 | 16 | 46 | 18 | 4 | 2
Days | 57.0 [20.0 to 218.0] | 75.0 [45.0 to 120.0] | 115.0 [59.0 to 174.0] | 102.0 [51.0 to 225.0] | 87.0 [52.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 64.5 [20.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

20. Secondary Outcome: Phase 1: PFS Per mRECIST v1.1
Description: According to mRECIST 1.1, PFS was defined as the length of time between the Baseline visit (Day 1) and the earlier of the participant's death or the first confirmed assessment of PD, as determined by investigator assessment of objective radiographic disease assessments. The response of target lesions was evaluated from the percentage change in the sum of the diameters of the viable portions (portions enhanced during the arterial phase).
Time Frame: up to approximately 44.7 months
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6
Days | 66.0 [48.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | NA [55.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 116.0 [64.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 88.0 [76.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 57.0 [29.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | NA [100.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 98.0 [52.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | NA [97.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 134.0 [53.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 128.0 [56.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | NA [46.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died.

21. Secondary Outcome: Phase 2: PFS Per mRECIST v1.1
Description: as for outcome 20
Time Frame: up to approximately 44.7 months
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 8 | 16 | 46 | 18 | 4 | 2
Days | 85.0 [20.0 to 218.0] | 105.0 [63.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 235.0 [129.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 168.0 [51.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 118.0 [52.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | NA [20.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died.

22. Secondary Outcome: Phase 1: Overall Survival
Description: Overall survival was defined as the interval between the Baseline visit (Day 1) and the date of death due to any cause.
Time Frame: up to approximately 44.7 months
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 5 | 4 | 4 | 4 | 8 | 3 | 6
Days | NA [76.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | NA [55.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | 253.0 [77.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 100.0 [76.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 289.5 [170.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 266.5 [100.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 588.0 [424.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 200.0 [97.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 425.0 [110.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 627.0 [128.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 229.5 [46.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

23. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival was defined as the interval between the Baseline visit (Day 1) and the date of death due to any cause.
Time Frame: up to approximately 44.7 months
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 8 | 16 | 46 | 18 | 4 | 2
Days | 290.5 [20.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 179.0 [75.0 to 404.0] | 491.0 [344.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 492.0 [92.0 to 733.0] | 485.0 [52.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 264.0 [20.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

24. Secondary Outcome: Phase 2: : Number of Participants With Any TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study medication.
Time Frame: up to approximately 27.4 months
Population: Phase 2 FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 8 | 16 | 46 | 18 | 4 | 2
Participants | 8. | 16 | 45 | 18 | 4 | 2

ADVERSE EVENTS:
Time Frame: up to approximately 27.4 months
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study medication, were monitored for at least 60 days after the last dose of study treatment or until the start of new anticancer therapy, whichever occurred first (up to 27.4 months). All-Cause Mortality was monitored for the duration of the study (up to 44.7 months).
Groups:
- Total: Total
Arm/Group | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg | Total
All-Cause Mortality (participants affected / at risk) | 2/4 | 2/4 | 4/5 | 3/4 | 4/5 | 4/4 | 3/4 | 4/4 | 5/8 | 2/3 | 6/6 | 6/8 | 12/16 | 25/46 | 11/18 | 3/4 | 2/2 | 98/145
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/4 | 3/5 | 2/4 | 2/5 | 1/4 | 2/4 | 2/4 | 3/8 | 1/3 | 2/6 | 3/8 | 11/16 | 19/46 | 10/18 | 2/4 | 1/2 | 68/145
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5 | 3/4 | 5/5 | 4/4 | 4/4 | 4/4 | 7/8 | 3/3 | 6/6 | 8/8 | 15/16 | 43/46 | 18/18 | 4/4 | 2/2 | 139/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W (N=4) | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W (N=4) | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W (N=5) | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W (N=4) | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W (N=5) | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W (N=4) | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W (N=4) | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W (N=4) | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W (N=8) | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W (N=3) | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab (N=6) | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg (N=8) | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg (N=16) | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg (N=46) | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg (N=18) | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg (N=4) | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg (N=2) | Total (N=145)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 8 (8)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary artery aneurysm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Group A: INCAGN01876 1.0 mg/kg Q2W + Nivolumab 240 mg Q2W (N=4) | Phase 1 Group A: INCAGN01876 3.0 mg/kg Q2W + Nivolumab 240 mg Q2W (N=4) | Phase 1 Group A: INCAGN01876 5.0 mg/kg Q2W + Nivolumab 240 mg Q2W (N=5) | Phase 1 Group A: INCAGN01876 10.0 mg/kg Q2W + Nivolumab 240 mg Q2W (N=4) | Phase 1 Group B: INCAGN01876 1.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W (N=5) | Phase 1 Group B: INCAGN01876 3.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W (N=4) | Phase 1 Group B: INCAGN01876 5.0 mg/kg Q2W, Then Nivolumab 240 mg Q2W (N=4) | Phase 1 Group C: INCAGN01876 1.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W (N=4) | Phase 1 Group C: INCAGN01876 3.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W (N=8) | Phase 1 Group C: INCAGN01876 5.0 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W (N=3) | Phase 1 Group D: INCAGN01876 + Nivolumab + Ipilimumab (N=6) | Phase 2 Group C2 PD-1/PD-L1 RM: INCAGN01876 300 mg + Ipilimumab 1 mg/kg (N=8) | Phase 2 Group F GC: INCAGN01876 300 mg + Nivolumab 240 mg (N=16) | Phase 2 Group F SCCHN INCAGN01876 300 mg + Nivolumab 240 mg (N=46) | Phase 2 Group F CC: INCAGN01876 300 mg + Nivolumab 240 mg (N=18) | Phase 2 Group F PD-1/PD-L1 RM: INCAGN01876 300 mg + Nivolumab 240 mg (N=4) | Phase 2 Group F Biopsy: INCAGN01876 300 mg + Nivolumab 240 mg (N=2) | Total (N=145)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 13 (13)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Allodynia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 7 (12) | 5 (6) | 0 (0) | 0 (0) | 25 (32)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 7 (7) | 1 (1) | 2 (2) | 0 (0) | 21 (22)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (11)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 7 (8)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 7 (10) | 2 (2) | 0 (0) | 0 (0) | 13 (17)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 16 (16)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder irritation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 7 (10)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Cestode infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clostridium test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 21 (22)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 12 (14) | 2 (3) | 0 (0) | 0 (0) | 27 (31)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 24 (24)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 6 (7) | 8 (11) | 8 (8) | 0 (0) | 0 (0) | 27 (31)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 13 (14)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 7 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 11 (11)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 23 (23)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 5 (6) | 15 (22) | 5 (5) | 1 (1) | 0 (0) | 40 (48)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (4)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 13 (16)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helminthic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 6 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 8 (9)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (9) | 1 (1) | 0 (0) | 0 (0) | 11 (13)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Inadequate analgesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 7 (7)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (11) | 0 (0) | 0 (0) | 0 (0) | 3 (11)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Medical device site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (11)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (6) | 2 (3) | 0 (0) | 3 (3) | 6 (7) | 7 (8) | 5 (5) | 1 (1) | 2 (2) | 35 (40)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 17 (17)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 8 (8)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 8 (8)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Penile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (4) | 3 (5) | 9 (9) | 7 (7) | 2 (3) | 0 (0) | 36 (41)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 15 (17)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 22 (26)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 6 (7)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (4)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 6 (8) | 1 (2) | 0 (0) | 0 (0) | 13 (17)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 9 (19)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (8) | 2 (3) | 0 (0) | 1 (1) | 21 (26)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT03126110/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03126110/SAP_001.pdf